CLINICAL TRIAL: NCT00743821
Title: Eye-Tracking Rapid Attention Computation
Acronym: Eye-TRAC
Status: Completed | Type: Observational
Sponsor: Brain Trauma Foundation (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, Jamshid Ghajar, M.D., Ph.D., President, Brain Trauma Foundation
Other Study IDs: PT075553; IRB Protocol #0211005884
Record Dates: First submitted 2008-08-28; First posted 2008-08-29 (Estimated); Last update posted 2014-05-07 (Estimated); Status verified 2014-05

CONDITIONS: Post Concussive Syndrome, Chronic
MeSH Terms: conditions — Post-Concussion Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- TBI Patients: Individuals who have suffered a mild traumatic brain injury and have persistent post-concussive symptoms (PCS)
- Normals: Individuals of comparable age and education who have not suffered a traumatic brain injury

SUMMARY:
The purpose of this study is to validate and refine a diagnostic device that can detect attention and memory deficits that result from mild traumatic brain injury (mTBI).

DETAILED DESCRIPTION:
The main goal of this project is the development of a military-ready, sensitive and rapid eye tracking diagnostic device for individuals with mild traumatic brain injury (mTBI). The device will also be tested for its efficacy in diagnosing fatigue and identifying aging effects. We will use a predictive visual tracking paradigm to dynamically capture the attentional state and correlate the subject's performance with the degree of disruption in the attention network caused by mTBI, aging and fatigue. The device will be tested for its diagnostic capabilities based on its selectivity, reliability, sensitivity and validity for individuals of varying ages (with and without mTBI) and in military personnel who have undergone 26 hours of sleep deprivation.

Testing will be conducted at two sites:

1. Civilians with mTBI; and civilians with adult attention deficit hyperactivity disorder will be tested by trained staff of the Brain Trauma Foundation (BTF) at Weill Cornell Medical College (WCMC) in New York City. The ages of the enrolled individuals will range between 18-55 years in order to examine aging effects.
2. Enrolled service members will be tested at the United States Army Research Institute of Environmental Medicine (USARIEM) in Natick, Massachusetts. These service members will be healthy volunteers without a history of mTBI. Some of these subjects will undergo 26 hours of sleep deprivation during which they will be tested at specific time points.

Our objectives are:

1. Prove that the eye-tracking concept can be brought from a successful laboratory device to a specific, reliable, selective, and valid diagnostic tool.

1.1. Test reliability by examining the test-retest reliability measures of EYE-TRAC;

1.2. Test selectivity by testing the ability to differentiating the effects of fatigue, aging, and mTBI on EYE-TRAC measures;

1.3. Test validity by determining the relationship between measures of attention and working memory based on the EYE-TRAC and validated measures of sustained attention and working memory;

1.4. Test specificity by measuring the spectrum of TBI injury using MRI-DTI and correlate with EYE-TRAC.

ELIGIBILITY:
Normals:

Inclusion Criteria:

* Healthy volunteer
* Education up to 12th grade

Exclusion Criteria:

* History of concussion or TBI
* Alcohol or substance abuse problems, neurological disorders, major psychiatric disorders (including ADHD or PTSD)
* Gross visual or hearing problems
* Pregnancy
* Metal in the body or any contraindications for MRI

TBI Patients:

Inclusion Criteria:

* Education up to 12th grade
* Persistent post concussive symptoms after an isolated incident of head injury with or without loss of consciousness between 3 months to 5 years prior to participation

Exclusion Criteria

* Prior history of seizures
* Pregnant woman
* Alcohol or substance abuse problems, neurological disorders, major psychiatric disorders (including ADHD or PTSD)
* Gross visual or hearing problems
* Any metal in the body or contraindications for MRI

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: TBI patients will be recruited from an outpatient TBI clinic Normals will be friends/family of TBI patients who have not suffered a TBI, as well as individuals recruited from the community
Sampling Method: Non-Probability Sample
Enrollment: 426 (Actual)
Dates: Start 2008-10; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jamshid Ghajar, M.D., Ph.D., Principal Investigator — Brain Trauma Foundation
Locations (1):
- Citigroup Imaging Center, Weill Medical College of Cornell University, New York, New York, United States